CLINICAL TRIAL: NCT03097068
Title: Analysis of Cytokines in Response to Treatment of Diabetic Macular Edema With 0.3mg Lucentis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vitreo-Retinal Associates, Michigan (Other)
Collaborators: Genentech, Inc. (Industry); Michigan State University (Other)
Responsible Party: Principal Investigator, Louis C Glazer, MD, Principal Investigator, Vitreo-Retinal Associates, Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ML39638
Record Dates: First submitted 2017-03-21; First posted 2017-03-31 (Actual); Results first posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 0.3 mg Lucentis (Experimental): Aqueous Humor sample post injection of 0.3 mg Lucentis
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: Lucentis — 0.3mg Lucentis
  Other Names: Aqueous Tap

SUMMARY:
The protocol will measure a number of cytokines in addition to vascular endothelial growth factor in response to 0.3mg Lucentis.

DETAILED DESCRIPTION:
Lucentis injections are the current standard of care for diabetic macular edema. The only deviation from the standard of care in the current protocol is an aqueous tap before the first Lucentis injection and the fourth Lucentis injection for diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus
* Best corrected visual acuity 20/32 - 20/320
* Diabetic macular edema involving the center of the macula
* Optical coherence tomography central subfield thickness of at least 250 microns

Exclusion Criteria:

* History of anti-vascular endothelial growth factor treatment in the past 12 months
* Any diabetic macular edema treatment in the past 4 months
* Heart attack, stroke, transient ischemic attack or acute congestive heart failure within 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vitreo-Retinal Associates, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.3 mg Lucentis
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 0.3 mg Lucentis
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 10
OCT Central Subfield Thickness [Mean (Standard Deviation); unit: microns] | 518.1 (257.19)

OUTCOME MEASURES:

1. Primary Outcome: Vascular Endothelial Growth Factor Levels
Description: An aqueous humor specimen was obtained at baseline and at 12 weeks to determine if the levels of VEGF had decreased with treatment.
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: pg/ml
Arm/Group | 0.3 mg Lucentis
Number analyzed (Participants) | 10
pg/ml | 73.46 [40.06 to 112.30]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | 0.3 mg Lucentis
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT03097068/Prot_SAP_000.pdf